CLINICAL TRIAL: NCT01254578
Title: A Phase 1 Study of Lenalidomide Maintenance Following Allogeneic Hematopoietic Cell Transplantation in Patients With Select High Risk Hematological Malignancies
Brief Title: Lenalidomide After Donor Bone Marrow Transplant in Treating Patients With High-Risk Hematologic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02551; NCI-2011-02551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 10079; OSU-10079; CDR0000688918; 2010C0069; OSU-2010C0069; OSU 10079 (Other: Ohio State University Comprehensive Cancer Center); 8305 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22.3;q23.3); MLLT3-KMT2A; Adult Acute Promyelocytic Leukemia With PML-RARA; Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-Cell Lymphoma; Alkylating Agent-Related Acute Myeloid Leukemia; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-Cell Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Hepatosplenic T-Cell Lymphoma; Intraocular Lymphoma; Lymphomatous Involvement of Non-Cutaneous Extranodal Site; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Nodal Marginal Zone Lymphoma; Post-Transplant Lymphoproliferative Disorder; Primary Cutaneous B-Cell Non-Hodgkin Lymphoma; Prolymphocytic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-Cell Leukemia/Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides and Sezary Syndrome; Recurrent Non-Hodgkin Lymphoma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Richter Syndrome; Small Intestinal Lymphoma; Splenic Marginal Zone Lymphoma; T-Cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Intraocular Lymphoma; Lymphoma, T-Cell; Leukemia, Prolymphocytic; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Lenalidomide

ARMS (1):
- Treatment (lenalidomide) (Experimental): Patients receive oral lenalidomide once daily on days 1-28. Courses repeat every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Patients undergo blood and bone marrow biopsies and aspirate collection at baseline and periodically during study for pharmacokinetic and pharmacodynamic studies. Buccal swab samples are also collected at baseline and analyzed for genetic polymorphisms.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given orally
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I clinical trial is studying the side effects and the best dose of lenalidomide after donor bone marrow transplant in treating patients with high-risk hematologic cancer. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximal-tolerable dose (MTD) of lenalidomide after allogeneic hematopoietic stem cell transplantation (AHSCT) in patients with advanced acute myeloid leukemia (AML), non-Hodgkin's lymphoma (NHL), or chronic lymphocytic leukemia (CLL).

II. Define the qualitative and quantitative toxicities of lenalidomide in regard to organ specificity, time course, predictability, and reversibility following AHSCT in these patients.

SECONDARY OBJECTIVES:

I. Determine the anti-tumor response in patients treated with lenalidomide after AHSCT when compared with historical controls.

II. Evaluate the plasma and cellular pharmacokinetics of lenalidomide in patients enrolled on this study and interactions with supportive agents such as calcineurin inhibitors.

III. Evaluate the frequency of acute and chronic graft-vs-host disease and graft failure in patients enrolled on this study.

IV. Prospectively assess the feasibility of administering an oral agent post-transplant as measured by efficiency of patients being registered to therapy early and also meeting eligibility criteria for lenalidomide treatment.

V. Perform pharmacodynamic studies following lenalidomide treatment including development of B, T, and myeloid cell chimerism; assessment of immune activation; cytokines; tumor cell expression of co-stimulatory molecules; development of anti-tumor antibodies and immunoglobulin recovery; and re-expression of microRNAs that may mediate lenalidomide anti-tumor effect.

OUTLINE: This is a multicenter, dose-escalation study. Patients are stratified according to diagnosis (high-risk acute myeloid leukemia vs non-Hodgkin lymphoma vs high-risk chronic lymphocytic leukemia, small lymphocytic lymphoma, or B-prolymphocytic leukemia).

Patients receive oral lenalidomide once daily on days 1-28. Courses repeat every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and bone marrow biopsies and aspirate collection at baseline and periodically during study for pharmacokinetic and pharmacodynamic studies. Buccal swab samples are also collected at baseline and analyzed for genetic polymorphisms.

After completion of study therapy, patients are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hematologic malignancy meeting 1 of the following criteria:

  * High-risk acute myeloid leukemia meeting 1 the following criteria:

    * First complete response (CR) and ≥ 60 years of age OR < 60 years of age with high-risk cytogenetics as defined by CALGB OR high-molecular risk and not eligible or willing to undergo myeloablative conditioning
    * Second or later complete remission
    * Not in remission but with < 5% blasts within 3 weeks of start of conditioning chemotherapy for allogeneic transplantation
    * Patients with a history of CNS involvement allowed provided disease is in remission at the time of transplantation
  * Patients with non-Hodgkin lymphoma who are candidates for allogeneic stem cell transplantation will be eligible; patients who have relapsed status post autologous transplantation are eligible as long as they demonstrate chemotherapy sensitive disease; patients with a history of CNS involvement are eligible if this aspect of the disease is in remission at the time of transplantation
  * High-risk chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or primary and secondary B-prolymphocytic leukemia (PLL) meeting 1 of the following criteria:

    * del(17p13.1) disease that has been treated (may have been given as consolidation therapy)
    * Less than PR to chemoimmunotherapy or relapsed within 2 years of treatment
    * Nucleoside analog refractory disease or disease that relapsed after two prior regimens
    * Patients with Richter (large cell) transformation allowed provided the large cell component of the disease is in remission (< 10% large cells in the bone marrow allowed)
* Patient has undergone an allogeneic stem cell transplantation using a reduced-intensity or non-myeloablative conditioning regimen within the past 60 days

  * At least 40% T-cell donor chimerism at day 30
* ECOG performance status 0-2 (Karnofsky 60-100%)
* Life expectancy > 3 months
* Myeloid engraftment with absolute neutrophil count > 1,000/μL and platelet count > 50,000/μL (after allogeneic hematopoietic stem cell transplantation [AHSCT])
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)

  * AST < 3 times ULN after AHSCT
* Creatinine clearance ≥ 50 mL/min in stratum 1 or ≥ 30 mL/min in stratum 2
* DLCO > 40% with no symptomatic pulmonary disease
* LVEF ≥ 30% by echocardiogram or MUGA
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must agree to use two acceptable methods of contraception (one highly effective method and one additional effective method) or practice abstinence for ≥ 28 days before, during, and ≥ 28 days after completing lenalidomide
* HIV negative
* No uncontrolled infection requiring intravenous therapy or poorly controlled diabetes mellitus
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No history of grade 3 or 4 graft-vs-host disease (GVHD)

  * If patient has acute GVHD grade 1 or 2, GVHD must be controlled and dose of oral prednisone or equivalent ≤ 20 mg per day (after AHSCT)
* More than 4 weeks since prior chemotherapy (excluding steroids), radiotherapy, or radioimmunoconjugate therapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2012-11-09 (Actual); Study Completion 2012-11-09 (Actual)

PRIMARY OUTCOMES:
MTD of lenalidomide after allogeneic hematopoietic stem cell transplantation graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 | Up to day 28

SECONDARY OUTCOMES:
Overall response in patients treated with lenalidomide according to the International Working Group (IWG) criteria | Up to day 365
  Estimated using exact binomial methods along with its confidence interval. The non-parametric Wilcoxon signed-rank procedure will be used to compare to baseline values for correlative studies.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Andritsos, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States